CLINICAL TRIAL: NCT01570348
Title: Allogeneic Hematopoietic Cell Transplantation for Patients With Treatment-Refractory Crohn's Disease: A Phase 2 Study
Brief Title: Crohn's Allogeneic Transplant Study
Acronym: CATS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Annual accrual goal not met
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2551.00; NCI-2011-03286 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2551; 2551.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; Allogeneic bone marrow transplantation; Hematopoietic cell transplantation
MeSH Terms: conditions — Crohn Disease | interventions — Cyclophosphamide; fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (allogeneic BMT) (Experimental): CONDITIONING THERAPY: Patients receive fludarabine phosphate IV over 30-60 minutes QD on days -6 to -2 and cyclophosphamide IV over 1-2 hours QD on days -6 and -5. Patients undergo total body irradiation on day -1.
  TRANSPLANTATION: Patients undergo donor BMT on day 0.
  IMMUNOSUPPRESSIVE THERAPY: Patients receive high-dose cyclophosphamide IV over 1-2 hours QD on days 3-4, tacrolimus IV daily or PO BID on days 5-180 with taper to day 365, and mycophenolate acid enteric coated or mycophenolate mofetil PO TID on days 0-35.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Drug: Mycophenolic Acid; Other: Quality-of-Life Assessment; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo allogeneic BMT
  Other Names: Allo BMT; Allogeneic BMT
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Drug: Mycophenolic Acid — Given PO
  Other Names: Acide mycophenolique; Acido micofenolico; Acidum mycophenolicum; Lilly-68618; Ly 68618; MPA; Myfortic
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase II trial studies how well giving a donor bone marrow transplant (BMT) works in treating patients with refractory Crohn's Disease. We will select patients with severe Crohn's Disease and active inflammation despite the best medical and surgical treatments. These patients must be healthy enough to undergo a transplantation procedure. They cannot have an active infection, and their heart, lungs, kidneys, and liver cannot be failing. The transplant procedure starts with chemotherapy and a small dose of radiation, to weaken a patient's immune system so that it will accept bone marrow cells from another person. After that other person's bone marrow cells are given to the patient, immune suppressive medicines are given to prevent the new cells from being rejected and to stop those cells from damaging the patient. After the new donor cells start to work, blood counts will rise and the new immune system will start to grow. During this time, there is a risk of infection. Antibiotics and anti-viral drugs will be given to prevent infection. When the new donor cells are well-established, immune suppressive medicines are discontinued. We will examine parts of the intestine that were inflamed before the start of the transplant procedure, to be sure the Crohn's Disease has disappeared after the transplant. Patients will be formally evaluated for Crohn's activity at around 100 days after transplant, and yearly after that for 5 years.

DETAILED DESCRIPTION:
BACKGROUND:

There is strong evidence for genetic susceptibility to Crohn's Disease (CD), with environmental factors interacting with genetic polymorphisms. Some patients remain refractory to the best available therapies. In patients with intestinal inflammation related to other genetic disorders, allogeneic hematopoietic cell transplantation has led to disappearance of inflammation, for example, in patients with IPEX (immune dysregulation, polyendocrinopathy, enteropathy, X-linked) and with a mutation in the Interleukin-10 receptor, characterized by a severe, early onset, fistulating colitis for which transplantation is the only therapy that offers benefit. Eleven patients with typical CD who achieved allogeneic donor chimerism after transplant had resolution of signs and symptoms of CD that was sustained for up to 15 years. These case series suggest that allogeneic transplantation has substantial potential to cure CD.

HYPOTHESIS AND SPECIFIC AIMS:

The hypothesis is: Allogeneic hematopoietic cell transplantation (HCT) can achieve sustained remissions in patients with refractory CD, and can be done safely. The specific aims are: 1) To evaluate the safety and efficacy of allogeneic HCT as treatment for refractory CD. 2) To evaluate treatment effect on CD activity/severity using the Crohn's Disease Activity Index (CDAI) and the Simple Endoscopic Score for CD (SES-CD). 3) To evaluate safety by scoring regimen-related toxicities, time to engraftment, infectious complications, acute and chronic Graft-versus-Host Disease (GVHD), and treatment-related mortality. 4) To evaluate the effect on quality of life.

METHODS:

This study is a prospective single-arm Phase II clinical trial that will enroll 12 patients.

PATIENT SELECTION: Patients will have documented CD (see eligibility criteria below); signs and symptoms that have failed to respond satisfactorily to medical and surgical therapies; active intestinal inflammation by endoscopy and histology, and CDAI >= 250 or need for total parenteral nutrition or recurrent inflammation after resection. Donors will be a Human Leukocyte Antigen (HLA)-matched sibling or unrelated donor.

ALLOGENEIC TRANSPLANT PROCEDURE: Patients will receive a reduced-intensity conditioning regimen of cyclophosphamide, fludarabine and low-dose Total Body Irradiation (TBI), a regimen that has been used successfully in patients receiving haploidentical allografts. Marrow will be used as the graft source to reduce the risk of GVHD. GVHD prophylaxis will consist of post-transplant high-dose cyclophosphamide followed by the combination of tacrolimus and enteric coated mycophenolic acid. Supportive care includes the use of N-acetyl cysteine infusions to reduce the risk of sinusoidal liver injury from cyclophosphamide; prophylaxis with ursodiol to prevent cholestatic liver disease; and antimicrobial drugs as prophylaxis and preemptive treatment for infections by bacteria, fungi, herpes viruses, and Pneumocystis jiroveci. Tissue and blood samples will be archived for future studies and evaluation of immune reconstitution at predefined intervals.

EFFICACY AND SAFETY ENDPOINTS: Safety and efficacy will be based on clinical assessments, laboratory testing, and gastrointestinal endoscopy and histology at baseline, at day 100 post-transplant, and yearly for 5 years. The primary endpoint is event-free survival at 1 year, defined as alive and free of active CD by endoscopy and biopsy. Transplant-related mortality is death occurring at any time after start of allogeneic HCT. Disease activity will be evaluated using CDAI. Quality of Life will be measured using the Short Inflammatory Bowel Disease Questionnaire.

RISKS AND POTENTIAL BENEFITS: The major risks include regimen-related toxicity, infections, graft rejection, and GVHD. Autologous stem cells will be reserved in case of graft rejection. Recent advances in transplant technique have substantially reduced the mortality risk. Balancing these risks is the potential for allogeneic transplant to effect sustained remissions and cures of CD.

PRIMARY OBJECTIVES:

I. The primary objective is to evaluate the safety and efficacy of HCT as treatment for refractory CD.

SECONDARY OBJECTIVES:

I. To evaluate treatment effect on CD activity and severity.

II. To evaluate safety of allogeneic HCT as determined by regimen-related toxicities, infectious complications, acute and chronic GVHD, treatment-related mortality, overall total mortality, and time to engraftment.

III. To evaluate the effect of allogeneic HCT on quality of life (QOL) in patients with severe refractory CD.

OUTLINE:

CONDITIONING THERAPY: Patients receive fludarabine phosphate intravenously (IV) over 30-60 minutes on days -6 to -2 and cyclophosphamide IV over 1-2 hours on days -6 and -5. Patients undergo 200 cGy of TBI on day -1.

TRANSPLANTATION: Patients undergo allogeneic BMT on day 0.

IMMUNOSUPPRESSIVE THERAPY: Patients receive high-dose cyclophosphamide IV over 1-2 hours on days 3-4, tacrolimus IV daily or orally (PO) twice daily (BID) on days 5-180 with taper to day 365, and mycophenolate acid enteric coated or mycophenolate mofetil PO three times daily (TID) on days 0-35.

After completion of conditioning therapy and infusion of donor bone marrow cells, patients are followed up at 1 month, 3 months, 12 months, and then yearly thereafter for up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CD established by referring physician(s) and confirmed by our review of the clinical presentation, clinical course, endoscopic and imaging findings, and histology of mucosal tissue specimens
* An adverse prognosis, documented by persistent signs and symptoms of CD that have failed to respond satisfactorily to medical and surgical therapies in the past, including but not limited to systemic immune suppressive drugs and biopharmaceuticals; to be considered as refractory to medical and surgical therapy, there must be clinical, endoscopic, and histologic evidence of active inflammatory Crohn's Disease that has either persisted or recurred despite exhaustive treatment with available pharmaceutical and surgical therapies; exhaustive treatment is defined as prior exposure to the following, without durable improvement:

  * Systemic glucocorticoids at or above a prednisone equivalent of 40 mg/day for at least 2 weeks, or until drug toxicity or intolerance develops
  * Methotrexate (25 mg per week for at least 3 months, or until drug toxicity or intolerance develops) and/or a thiopurine antimetabolite (either 2.5 mg/kg azathioprine or 1.5 mg/kg 6-mercaptopurine in patients homozygous wild-type for the thiopurine-S-methyltransferase [TPMT] gene, or either 1.5 mg/kg azathioprine or 1 mg/kg 6-mercaptopurine in patients heterozygous for TPMT, or doses of these drugs capable of producing a 6-thioguanine nucleotide level of 230-400 without producing a 6-methylmercaptopurine nucleotide level above 5700 for at least 3 months, or until drug allergy, intolerance or toxicity develops); if a patient is homozygous mutant for the TPMT gene, thiopurines would be contraindicated and their use would not be a requirement for enrollment in this protocol
  * Use of at least two anti-tumor necrosis factor (TNF)-alpha therapies, that is, infliximab (at least 5 mg/kg every 8 weeks for at least 3 months, or until drug allergy, toxicity or intolerance or anti-infliximab antibodies develop) and/or adalimumab (at least 40 mg subcutaneously [SQ] every 2 weeks for at least 3 months, or until drug allergy, toxicity or intolerance develops) and/or certolizumab pegol (at least 400 mg SQ every 4 weeks for at least 3 months, or until drug allergy, toxicity or intolerance develops)
  * Due to the serious risk of progressive multifocal leukoencephalopathy (PML) and the reluctance of some patients to agree to therapy that carries such risk, prior exposure to natalizumab is not required to meet the definition of exhaustive pharmaceutical treatment; neither will use of natalizumab among patients who are John Cunningham (JC) virus antibody seronegative be an exclusionary criterion
  * Exhaustive surgical treatment will be defined as indicated operations for complications of Crohn's Disease up to the point where the risks of surgery (for example, mortality or post-operative morbidity such as short bowel syndrome or extensive adhesions with high risk for inadvertent enterotomy) are deemed by patients and their physicians to be unacceptably high; indicated operations for complications of Crohn's Disease include, but are not limited to, surgical resection of involved intestine, stricturoplasty, drainage, curettage, or adhesiolysis of tissues affected by Crohn's disease
  * Exposure of patients to investigational drug therapies for Crohn's Disease, that is, to drugs that are not Food and Drug Administration (FDA) approved for this indication, will not be a criterion for either inclusion or exclusion
* Endoscopic and histologic evidence of active intestinal inflammation consistent with CD; in the event that the involved mucosa cannot be readily reached by endoscopic biopsy, an imaging test that shows typical changes of CD in the intestinal tract will suffice as evidence of active intestinal inflammation; the presence of intestinal stomas does not exclude the patient from study
* Severe CD as defined by one of the following:

  * CDAI >= 250
  * Need for total parenteral nutrition to maintain weight
  * Recurrent intestinal inflammation caused by CD following surgical resection
* Identification of a HLA-matched hematopoietic cell donor without a history of a disorder that can be transmitted by hematopoietic cells, including but not limited to inflammatory bowel disease, and without nucleotide-binding oligomerization domain containing 2 (NOD2) mutations in the case of a HLA matched sibling
* DONORS will be a HLA-identical sibling or HLA-matched unrelated donor; unrelated donors are required to be matched by high resolution allele level typing for HLA-A, B, C and DRB1 and intermediate resolution Sequence Specific Oligonucleotide Probes (SSOP), identifying alleles in groups of related families historically defined as antigens for DQB1; an unrelated donor is considered matched if patient and donor share HLA-A, B, C alleles with identical sequences at exons 2 and 3, DRB1 alleles with identical sequences at exon 2, and DQB1 results that include the same allele groups
* DONORS will have the ability to understand and the willingness to sign a written informed consent document for bone marrow harvest.

Exclusion Criteria:

* A current complication of CD that would jeopardize survival after hematopoietic cell transplantation, including but not limited to the following:

  * Abscess, phlegmon, necrotizing skin lesion, or inflammatory fistula
  * Intestinal fibrotic stricture and intestinal obstruction
  * Uncontrolled mucosal, organ, or systemic infection with a bacterial, viral, fungal, or parasitic organism
  * Sclerosing cholangitis
* History of progressive multifocal leukoencephalopathy
* Organ dysfunction or disease that would jeopardize survival after hematopoietic cell transplantation, including but not limited to the following:

  * Renal insufficiency as defined by an estimated glomerular filtration rate (GFR) < 60 mL/minute
  * Cardiac dysfunction as defined by symptomatic coronary artery disease, congestive heart failure, valvular heart disease, cardiomyopathy, uncontrolled arrhythmia(s), or left ventricular ejection fraction < 50%
  * Pulmonary dysfunction that poses a risk of mortality after transplant, defined as pulmonary disease-moderate, using pre-transplant pulmonary function testing per the Fred Hutchinson Cancer Research Center (FHCRC) Standard Practice Manual
  * Necroinflammatory or fibrotic liver disease with evidence of liver dysfunction, including but not limited to jaundice, hepatic encephalopathy, or portal hypertension
  * Marrow dysfunction that poses a risk of peri-transplant mortality, defined as an absolute neutrophil count or lymphocyte count below the lower limit of normal, or a platelet count below 50,000/mm^3
  * Poorly controlled hypertension despite appropriate therapy, defined as a diastolic blood pressure greater than 90 mm Hg while on therapy
  * Neurologic dysfunction that affects activities of daily living and medical care
  * Poorly controlled diabetes mellitus, defined as persistent hyperglycemia despite therapy or recurrent hypoglycemia while on therapy
  * Extreme protein-calorie malnutrition defined by body mass index < 18 kg/m^2 and unintentional weight loss (3 kg in the last month or 6 kg in the last 6 months)
* Pregnancy
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following transplant
* History of smoking either tobacco or other herbal products in the last 3 months
* Human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) seropositivity
* Patients whose life expectancy is severely limited by illness other than CD
* Untreated psychiatric illness, including drug/alcohol abuse, that would compromise compliance
* Inability to give voluntary informed consent or obtain a parent or guardian's informed consent
* Demonstrated lack of compliance with prior medical care
* History of a malignancy, excluding adequately treated squamous cell skin cancer, basal cell carcinoma, and carcinoma in situ
* Hematopoietic cell transplant-co-morbidity Index greater than 2
* DONOR: Identical twin
* DONOR: Pregnant or lactating females
* DONOR: HIV seropositivity or presence of HBV deoxyribonucleic acid (DNA) or HCV ribonucleic acid (RNA) in the serum
* DONOR: Current serious systemic illness including uncontrolled infections
* DONOR: Malignancy within 10 years prior to donation of marrow, excluding adequately treated squamous cell skin cancer and basal cell carcinoma; treatment must have been completed (with the exception of hormonal therapy for breast cancer) with cure/remission status verified for at least 10 years at time of marrow harvest
* DONOR: History of or symptoms consistent with inflammatory bowel disease or a serious autoimmune disorder
* DONOR: Homozygous NOD2 mutation
* DONOR: History of a serious disease or disorder that could be adoptively transferred by infusion of donor hematopoietic cells
* DONOR: Failure to meet institutional criteria for donation as described in the Standard Practice Guidelines

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2012-07-17 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Georges, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] McDonald GB, Landsverk OJB, McGovern DPB, Aasebo A, Paulsen V, Haritunians T, Reims HM, McLaughlin BM, Zisman T, Li D, Elholm ETMM, Jahnsen FL, Georges GE, Gedde-Dahl T. Allogeneic bone marrow transplantation for patients with treatment-refractory Crohn's Disease. Heliyon. 2024 Jan 3;10(1):e24026. doi: 10.1016/j.heliyon.2024.e24026. eCollection 2024 Jan 15. PMID 38283244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited 7/2012 and 8/2015 via website (www.CATS-FHCRC.org). Over 700 completed questionnaires, >150 were deemed potentially eligible. 15 completed records reviewed and invited for in-depth screening for eligibility. Two study participants were enrolled.
Groups:
- Treatment (Allogeneic BMT): CONDITIONING THERAPY: Patients receive fludarabine phosphate IV over 30-60 minutes QD on days -6 to -2 and cyclophosphamide IV over 1-2 hours QD on days -6 and -5. Patients undergo total body irradiation on day -1.
  TRANSPLANTATION: Patients undergo donor BMT on day 0.
  IMMUNOSUPPRESSIVE THERAPY: Patients receive high-dose cyclophosphamide IV over 1-2 hours QD on days 3-4, tacrolimus IV daily or PO BID on days 5-180 with taper to day 365, and mycophenolate acid enteric coated or mycophenolate mofetil PO TID on days 0-35.
  Allogeneic Bone Marrow Transplantation: Undergo allogeneic BMT
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Mycophenolic Acid: Given PO
  Quality-of-Life Assessment: Ancillary studies
  Tacrolimus: Given IV or PO
  Total-Body Irradiation: Undergo TBI
Period: Overall Study
Arm/Group | Treatment (Allogeneic BMT)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Norway | 1
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: Defined as alive and free of active CD. Described graphically using a Kaplan-Meier estimate. Generated with confidence intervals using Greenwood's formula to calculate the standard error. Estimated with exact 90% confidence intervals.
Time Frame: At 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Participants | 1

2. Secondary Outcome: Development of Infectious Complications
Description: The incidence of definite and probable viral, fungal and bacterial infections will be tabulated for each patient.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Participants | 1

3. Secondary Outcome: Disease Activity
Description: Evaluated using a standardized tool for evaluating CD (CDAI).
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Participants | 0

4. Secondary Outcome: EFS
Description: Described graphically using a Kaplan-Meier estimate. Generated with confidence intervals using Greenwood's formula to calculate the standard error. Estimated with exact 90% confidence intervals.
Time Frame: Up to 5 years post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Participants | 1

5. Secondary Outcome: Incidence and Severity of GVHD
Description: The grading of acute and chronic GVHD will follow previously published guidelines but will also include capture of symptoms and characterization of alternative causes. The highest level of organ abnormalities, the etiologies contributing to the abnormalities and biopsy results pertaining to GVHD will be identified. Since both GVHD and CD involve the gastrointestinal tract, all diagnostic biopsies of these organs will be reviewed by pathologists experienced in the diagnosis of GVHD and IBD, respectively.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Participants | 1

6. Secondary Outcome: Incidence of Disease-modifying Drugs for CD Initiated Post-transplant
Description: Includes the administration of any therapy (drugs, biologics, or any other treatments) clearly given as immunomodulatory therapy for underlying CD.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Participants | 0

7. Secondary Outcome: Incidence of Graft Rejection
Description: Engraftment is defined as achieving > 5% donor peripheral blood CD3 T cell chimerism by day 84 after HCT. Primary graft failure is defined as a donor peripheral blood CD3 T cell chimerism peak of < 5% by Day 84 post-HCT. Secondary graft failure is defined as documented engraftment followed by loss of the graft with donor peripheral blood CD3 T cell chimerism < 5% as demonstrated by a chimerism assay.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Participants | 0

8. Secondary Outcome: Overall Survival
Description: Characterized by the event rates as functions of all patients enrolled and at risk of the event, with exact confidence intervals.
Time Frame: Time of treatment assignment until death due to any cause, assessed up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Participants | 1

9. Secondary Outcome: Quality of Life Measured Using the Previously Validated Short Inflammatory Bowel Disease Questionnaire
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Participants | 0

10. Secondary Outcome: Regimen-related Toxicity Graded According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4
Description: Characterized by the rates of reportable events as functions of all patients enrolled and at risk of the event, with exact confidence intervals. With the exception of adverse events (AEs) that are universal and expected following conditioning therapy, all reportable AEs will be tabulated for each patient from the time that the subject starts mobilization of hematopoietic cells until day +365 after transplant.
Time Frame: Up to 1 year post-BMT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Participants | 1

11. Secondary Outcome: Treatment-related Mortality (TRM)
Description: A stopping rule will be imposed for TRM occurring within one year of transplant. The study will be stopped if at any point there is moderately strong evidence that the rate of TRM exceeds 10%. Moderately strong evidence will be taken to mean that the lower bound of a one-sided 80% confidence interval for the true rate of TRM is above 10%.
Time Frame: Time from BMT to death definitely or probably resulting from treatment, assessed up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Allogeneic BMT)
Number analyzed (Participants) | 2
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events collected from mobilization start until day +365 after allogeneic HCT or patient withdraws from the study. After HCT- day +100, grades 3, 4 and 5 adverse events will be captured, exception outlined in Appendix J. Grades 3 and 4 adverse events in CD involved organs only if they represent a significant change from baseline status. Day+100- +365 only Grades 4 and 5.
Arm/Group | Treatment (Allogeneic BMT)
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Allogeneic BMT) (N=2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Allogeneic BMT) (N=2)
thromboembolotic event (Vascular disorders) | 1 (1)
CMV Reactivation (Infections and infestations) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Femoral neck stress fracture (Injury, poisoning and procedural complications) | 1 (1)
metapneumovirus pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Respiratoroy failure (Respiratory, thoracic and mediastinal disorders) | 1 (3)
acute kidney injury (Renal and urinary disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
GI bleed/dirrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT01570348/Prot_SAP_000.pdf